CLINICAL TRIAL: NCT03213860
Title: The Effect of Night Eye Mask on Post-operative Pain in Cardiac Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pain & Sleep
Record Dates: First submitted 2017-07-02; First posted 2017-07-11 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Sleep Deprivation; Postoperative Pain
MeSH Terms: conditions — Sleep Deprivation; Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: While it is not possible to blind participants and clinical staff to the assigned interventions, the assessments will be undertaken by a researcher blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eye mask (Active Comparator)
  Interventions: Other: Flight Eye-masks; Dreaming, Zhuji City, Zhejiang, China
- Control (No Intervention)

INTERVENTIONS:
Other: Flight Eye-masks; Dreaming, Zhuji City, Zhejiang, China — The experimental group will receive protective devices Single use eye masks during nocturnal sleep (Flight Eye-masks; Dreaming, Zhuji City, Zhejiang, China). The caregiver will explain to them that they should wear eye masks during their stay in ICU to ensure rest and instructed patients to use them properly. During the ICU stay, ICU nurses will assist patients with wearing eye masks from 9:00 pm to 7:00 am the next morning.
  Arms: eye mask

SUMMARY:
Environmental factors such as noise and light have been cited as important causes of sleep deprivation in Intensive care unit (ICU) patients. Previous studies demonstrated a hyperalgesic alteration in pain perception following a controlled sleep deprivation protocol. Another studies indicated that using eye masks can improve REM sleep in healthy subjects in simulated ICU environment, and improve sleep quality in ICU patients. This study aimed to determine the effects of using eye masks on sleep and thus on pain quality in postoperative cardiac surgery patients in ICU.

ELIGIBILITY:
Inclusion Criteria:

* (1) age ≧18 years; (2) no history of neurological or psychiatric disorders; (3) ability of patients to communicate verbally and understand the sleep questionnaires administered in the ICU; (3) length of ICU stay ≥48 hours; (4) Glasgow coma score (GCS) >8 in the first to third day. Postoperative Extubation of MV within few hour (before the time of 9 pm for postoperative patients.

Exclusion Criteria:

* Patients over age 65 were excluded from the study because of potential age-related differences in sleep. Patients reporting frequent nighttime awakenings, snoring, or chronic use of benzodiazepines or opioids were excluded because of potential confounding influences of these factors on postoperative sleep, pain, or opioid requirement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 3 postoperative days
  visual analogue scale will be used. ranging from 0 mm (no pain) to 100 mm (worst pain imaginable).

SECONDARY OUTCOMES:
Quality of sleep | 3 postoperative days
  the Arabic version of the Richards-Campbell Sleep Questionnaire (RCSQ)The five-point RCSQ was designed to evaluate different aspects of night-time sleep, including: (1) depth; (2) latency (time to fall asleep); (3) number of awakenings; (4) efficiency (percent of time awake), and (5) quality. Each item was scored using a 100-mm visual-analogue scale (VAS), which ranged from 0 mm (worst sleep) to 100 mm (optimal sleep). Total score was calculated by dividing the sum of all scores by five. The RCSQ was administered by the researcher daily, at 7:00am every morning.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No